CLINICAL TRIAL: NCT00715728
Title: Efficacy of a New Intraoperative Resistive Warming Device
Brief Title: Efficacy of Warming Device During Surgery
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: IRWS
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2017-04

CONDITIONS: Surgery
Keywords: Plastic surgery; Warming; Core temperature; Bair Hugger; Hot Dog heating system

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Bair Hugger: Intraoperative warming with Bair Hugger forced air system
  Interventions: Device: Intraoperative warming with Bair Hugger forced air system
- 2: Hot Dog: Intraoperative warming with Hot Dog resistive heating system
  Interventions: Device: Intraoperative warming with Hotdog resistive heating system

INTERVENTIONS:
Device: Intraoperative warming with Bair Hugger forced air system — Intraoperative warming with Bair Hugger forced air system
  Groups: 1: Bair Hugger
Device: Intraoperative warming with Hotdog resistive heating system — Intraoperative warming with Hotdog resistive heating system
  Groups: 2: Hot Dog

SUMMARY:
This study will test the hypothesis that an electric heating device, the Hot Dog warming system is as effective as the Bair Hugger forced air heating system.

DETAILED DESCRIPTION:
Subjects undergoing major plastic surgery lasting approximately 5 hours will be randomized to either the Hot Dog resistive heating system or the Bair Hugger forced air heating system. Core temperature will be measured using a distal esophagus and mean skin temperature. Warming will continue until the subjects' core temperature reaches 37°C. Subsequent temperature will be adjusted as clinically necessary. Data will be recorded at 15 minute intervals. Core temperature will be first measured after intubation when the esophageal temperature probe is inserted. The primary outcome will be the rate of core rewarming over the range of 35°C to 37°C.

ELIGIBILITY:
Inclusion Criteria:

* Plastic surgery lasting approximately 5 hours
* Subjects over the age of 18 years
* Patient signed Informed Consent

Exclusion Criteria:

* Plastic surgery lasting less than 5 hours
* Individuals under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major plastic surgery lasting approximately 5 hours.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Plattner, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Vienna General Hospital/University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intra-operative Rewarming With Bair Hugger Heating: Intra-operative rewarming with Bair Hugger heating system
- Intraoperative Rewarming With Hot Dog Resistive Heating: Intraoperative rewarming with Hot Dog resistive heating system
Period: Overall Study
Arm/Group | Intra-operative Rewarming With Bair Hugger Heating | Intraoperative Rewarming With Hot Dog Resistive Heating
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bair Hugger Forced Air System: Patients were warmed with the Bair Hugger forced air system during surgery.
- Hot Dog Resistive Heating System: Patients were warmed with the Hot Dog resistive heating system during surgery.
- Total: Total of all reporting groups
Arm/Group | Bair Hugger Forced Air System | Hot Dog Resistive Heating System | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 12 | 8 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Core Rewarming Over the Range From 35°C to 37°C.
Description: The primary outcome was the rewarming rate during active heating over a core temperature range from 35°C to 37°C.
Time Frame: Until the end of surgery, up to 5 hour
Measure: Mean (Standard Error); unit: degrees Celcius / hr
Groups:
- Intra-operative Rewarming With Hot Dog: Intraoperative warming with Bair Hugger forced air system
- Intra-operative Rewarming With Forced-air Heating: Intraoperative warming with forced-air heating system
Arm/Group | Intra-operative Rewarming With Hot Dog | Intra-operative Rewarming With Forced-air Heating
Number analyzed (Participants) | 14 | 14
degrees Celcius / hr | .24 (.025) | .49 (.027)
Statistical Analysis 1: Comparison: Intra-operative Rewarming With Hot Dog vs Intra-operative Rewarming With Forced-air Heating; A total of 46 patients (23 per group) were needed to have 90% power to demonstrate equivalence of the two warming methods on final intra-operative temperature at the 0.05 significance level using the 2 one-tailed tests equivalence testing technique and an equivalence region of 0.5 degrees C per hour, assuming a SD of 0.5 degrees C/hour for each group and zero true difference; Test type: Equivalence — Our primary outcome was the rate of core rewarming during the surgery. Groups were compared on mean rewarming rate in a linear mixed effects regression model with within-subject change of core temperature over time as random effect. Using those model results, equivalence on the mean rate of rewarming for the resistive and warm air systems was assessed with the 2 one-tailed tests equivalence testing approach and equivalence delta of 0.2 degrees C/hours; p = 0.91, t-test, 1 sided — Two 1-tailed tests were conducted. P-value for lower delta was 0.91. Equivalence will be claimed if p-values for upper and lower delta are both lower than 0.05 ⁄ 2 = 0.025; Two 1-tailed tests were conducted to assess equivalence. See " Type of Statistical Test"
Statistical Analysis 2: Comparison: Intra-operative Rewarming With Hot Dog vs Intra-operative Rewarming With Forced-air Heating; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Intraoperative Time Weighted Average Core Temperature
Description: Temperatures during surgery were recorded at 15-min intervals and summarize as time weighted average (TWA) for each patient. The unit of TWA-temperature is °C.
Time Frame: Until the end of surgery, up to 5 hour
Population: Medical University of Vienna adults having major maxillary-facial reconstructive surgery expected to last about 5 h. Most had pectoral flap reconstructions after extensive cancer debridement. We did not study patients with Reynaud's disease, thyroid dysfunction, insulin-dependent diabetes mellitus, or who were of ASA physical status > 3.
Measure: Mean (Standard Error); unit: degrees as measured in Celcius
Groups:
- Intraoperative Warming With Bair Hugger Forced Air System: Intraoperative temperature warming with Bair Hugger forced air system
- Intraoperative Warming With Hot Dog Resistive Heating System: Intraoperative temperature warming with Hot Dog resistive heating system
Arm/Group | Intraoperative Warming With Bair Hugger Forced Air System | Intraoperative Warming With Hot Dog Resistive Heating System
Number analyzed (Participants) | 14 | 14
degrees as measured in Celcius | 36.24 (0.27) | 36.12 (0.25)
Statistical Analysis 1: Comparison: Intraoperative Warming With Bair Hugger Forced Air System vs Intraoperative Warming With Hot Dog Resistive Heating System; Null hypothesis is the Hot dog resistive heating system is inferior to the Bair Hugger forced air system. Mean difference (95% CI) of the intraoperative TWA temperature between the groups (resistive heating versus forced-air) will be adjusting for preoperative oral temperature and ASA physical status; Test type: Non-Inferiority — The non-inferiority margin is defined as 0.5 °C. Non-inferiority at the 0.025 significance level will be claimed if the lower limit of the 95% confidence interval is higher than the -0.5 °C; p = 0.018, t-test, 1 sided — P-value was adjusted for preoperative oral temperature and ASA physical status; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.37 to 0.14] — Non-inferiority will be established, at the 0.025 significance level, if the lower limit of a 95% confidence interval for the difference is above -0.5 °C

ADVERSE EVENTS:
Time Frame: From the beginning of the surgery until the end of surgery, up to 24 hour.
Description: Serious adverse events.
Arm/Group | Bair Hugger Forced Air System | Hot Dog Resistive Heating System
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
Unable to evaluate safety with small sample size. Smaller-than-expected sample size had enough power but confidence intervals for treatment effect wider than desired.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No